CLINICAL TRIAL: NCT06646263
Title: Cellular Immune Responses in Triple-negative Breast Cancer - High Throughput Immunogenetic Studies
Status: Enrolling by invitation | Type: Observational
Sponsor: Institute of Applied Biosciences (Other)
Collaborators: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: INAB017635
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Triple Negative Breast Cancer
Keywords: T cells; Tumor-infiltrating lymphocytes; Next-generation sequencing; T cell receptor; Spatial transcriptomics; Neoepitopes; TR beta chain; TRb clonotypes; TRb gene repertoire; Cellular immunity
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biospecimens include FFPE tumor samples and peripheral blood (PB) samples derived from TNBC patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This project introduces a novel methodology for the in-depth immunogenetic characterization of the TR gene repertoire in solid tumors, holding the promise to offer unprecedented insights into the TR anti-tumor specificity and the prognostic/predictive value of TR gene repertoire signatures.

DETAILED DESCRIPTION:
The goal of this observational study is to address the role of T cells in the tumor microenvironment of TNBC.

In detail, this study aims to:

(i) explore the immunogenetic characteristics of the TR gene repertoire as informative prognostic/predictive biomarkers in TNBC (ii) identify immunogenic neoepitopes arising from common tumor-specific non-synonymous gene mutations, as well as the corresponding neoepitope-specific T cells (iii) describe, in single-cell resolution, the spatial organization of the intricate crosstalk between tumor cells and neoepitope specific-T cells, and (iv) delineate the functional properties of T cells within the TME.

All the experimental results, regarding the TR repertoire features and the spatial organization of the TME, will be correlated with clinical outcome measurements (e.g. overall survival, progression time), which are available from the detailed patients medical record.

ELIGIBILITY:
Inclusion Criteria:

- Confirmed TNBC diagnosis

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study group includes patients diagnosed with TNBC. Each patient provided written informed consent, and paired samples of peripheral blood (PB) and tumor tissue were obtained at the time of diagnosis and before initiating any treatment. The selection of patients will be meticulously carried out by the PI and team members based on comprehensive clinical records, including clinicobiological characteristics. Further refinement of the study group will be contingent upon sample availability and the quality of biological material.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
T cell receptor profiling as a potential biomarker in Triple-Negative Breast Cancer | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Applied Biosciences, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided